CLINICAL TRIAL: NCT05425316
Title: Analysis of Acoustic, Lexical, and Syntactic Speech Features in Hepatic Encephalopathy
Brief Title: Speech in Hepatic Encephalopathy (HE)
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Winterlight Labs (Industry)
Responsible Party: Principal Investigator, Patricia Bloom, Assistant Professor, University of Michigan
Other Study IDs: HUM00191626
Record Dates: First submitted 2022-05-14; First posted 2022-06-21 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Cirrhosis: This group will be composed of 200 patients with cirrhosis. Patients will be enrolled regardless of compensated vs. decompensated status, prior history of HE, Model for End Stage Liver Disease (MELD), and cirrhosis etiology.
  Interventions: Behavioral: Home Recordings; Behavioral: In-patient Recordings; Behavioral: Same-Day Study Visit - Regular Appointment; Behavioral: Same-Day Study Visit - Procedure; Behavioral: Phone Call Follow-up Visits
- Patients without Cirrhosis: This group will be composed of 50 patients without cirrhosis to act as controls. They will have been found on Fibroscan to not have significant fibrosis.
  Interventions: Behavioral: Home Recordings; Behavioral: Same-Day Study Visit - Regular Appointment

INTERVENTIONS:
Behavioral: Home Recordings — If patients are willing to download the Winterlight application to their personal iOS devices this will be done at study visit 1. The application will send a notification to the patient once per month, requesting that they perform a paragraph reading task, a picture description task, and an animal naming task.
Behavioral: In-patient Recordings — If patients are admitted to UM hospital for suspected or confirmed OHE, with patient assent, physician study staff will assist the patient in recording a paragraph reading task, a picture description task, and an animal naming task.
  Groups: Patients with Cirrhosis
Behavioral: Same-Day Study Visit - Regular Appointment — Staff will call patients in anticipation of in-person regular visits to set up a same-day study visit. Patients will record the three speech tasks at this time.
Behavioral: Same-Day Study Visit - Procedure — Staff will call patients in anticipation of in-person procedure visits to set up a same-day study visit, prior to procedure if sedation is planned. Patients will record the three speech tasks at this time.
  Groups: Patients with Cirrhosis
Behavioral: Phone Call Follow-up Visits — Non-physician study staff will call the patients every 3 months and, using a phone script, will ask them survey questions about their hepatic health.
  Groups: Patients with Cirrhosis

SUMMARY:
This is an observational study that will test the clinical significance of speech features in patients with cirrhosis. It aims to assess if speech is associated with cognitive function at baseline, if speech predicts changes in cognition, and if speech predicts future events of hepatic encephalopathy (cirrhosis-related confusion), as well as to assess the dynamics of speech over time, especially with episodes of overt hepatic encephalopathy (OHE) and treatment interventions.

ELIGIBILITY:
Inclusion Criteria for Patients with Cirrhosis:

* Cirrhosis, as diagnosed by imaging, elastography, biopsy, or decompensation
* Able to provide informed consent in English

Exclusion Criteria for Patients with Cirrhosis:

* Neurodegenerative disorder (other than hepatic encephalopathy) including Alzheimer's disease and dementia
* Prior stroke or Transischemic Attack (TIA)
* English not primary language for communication

Inclusion Criteria for Patients without Cirrhosis:

* Able to provide informed consent in English
* Fibroscan with stiffness <7 kPa

Exclusion Criteria for Patients without Cirrhosis:

* Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) >5 times the upper limit of normal in the last year
* History of cirrhosis by imaging or histology or clinical decompensation
* Neurodegenerative disorder (other than hepatic encephalopathy) including Alzheimer's disease and dementia
* Prior stroke or TIA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of adult outpatients who are evaluated at the University of Michigan Hepatology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Change in Psychometric Hepatic Encephalopathy Score (PHES) from Baseline to 6 Months | 6 Months
  A well-validated pen-and-paper neurocognitive assessment tool to identify minimal Hepatic Encephalopathy (HE). Scores range from -15 to +5; values farther from 0 (normalized average) represent more significant deviation from the norm. Positive scores indicate better performance.
Change in Psychometric Hepatic Encephalopathy Score (PHES) from Baseline to 12 Months | 12 Months
  A well-validated pen-and-paper neurocognitive assessment tool to identify minimal Hepatic Encephalopathy (HE). Scores range from -15 to +5; values farther from 0 (normalized average) represent more significant deviation from the norm. Positive scores indicate better performance.
Speech Assessments | 12 Months
  Recorded speech tasks comprising 3 sections: paragraph reading test, picture description test, and animal naming test.
Time to Overt Hepatic Encephalopathy (HE) | 12 Months
  Patient-reported HE episodes and HE episodes resulting in patient admission to University of Michigan hospital. Information collected includes: Date of symptom onset, duration of HE episode, and changes to medications.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bloom, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hepatology and Transplant Clinic, Ann Arbor, Michigan, United States